CLINICAL TRIAL: NCT02077816
Title: Using Non-contact Infrared Thermometry to Detection of Central Venous Catheter Related Infection.
Brief Title: Using a Infrared Thermometer to the Early Detection of Catheter Related Infections
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Julio Sergio Marchini, Full Professor of Internal Medicine Department at Ribeirão Preto Medical School, University of Sao Paulo
Other Study IDs: HCRP 12632/2010; CAAE - 0444.0.004.000-10 (Registry Identifier: Sistema Nacional de Informações sobre Ética em Pesquisa)
Record Dates: First submitted 2014-03-02; First posted 2014-03-04 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-03

CONDITIONS: Infection
Keywords: body temperature; Thermometry; Infrared Rays; catheter related infection
MeSH Terms: conditions — Infections; Catheter-Related Infections

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Central venous catheter: Inpatients with CVC for medical care.

SUMMARY:
This is a pilot study which aims to show the temperatures measured on body surface with an infrared thermometer on inpatients who need a central venous catheter (CVC) for medical care. Because the local temperature could be altered, at least during local infectious processes, seems to be reasonable to think that this approach could be helpful to its early diagnosis.

DETAILED DESCRIPTION:
By convenience sampling, it was expected that during 4 months, a minimum of 30 inpatients of the metabolic, clinical or intensive care wards, at the Clinical Hospital of Ribeirão Preto Medical School, São Paulo, Brazil, would have their data collected

ELIGIBILITY:
Inclusion Criteria:

* Need of a central venous catheter for medical care.
* Be an inpatient of the metabolic, clinical or intensive care wards

Exclusion Criteria:

* Be in treatment course of a catheter related infection.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Inpatient of the metabolic, clinical or intensive care wards with a CVC for medical care.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2011-08; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Body temperature measured with a non-contact infrared thermometer. | 15 minutes after bath, mobilization or warm or cold compresses
  It was used a non-contact forehead infrared thermometer, model IR200® (Extech, USA). Fifteen minutes after bath, mobilization or warm or cold compresses, 3 measurements were obtained at the following sites: 1) close to CVC insertion, 2) at the equivalent contralateral site of CVC and 3) at the forehead. The variables values will be displayed in form of descriptive statistics (mean, standard deviation, standard error, proportions of the observations, confidence intervals) according to: sex, central venous catheter type (guide wire or port-a-cath), location of insertion, reason of the central venous catheter indication (like parenteral nutrition or antibiotics), number of catheter lumens and age. Also, the mean differences between the three locations measured will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Júlio S Marchini, Ph.D, Principal Investigator — Ribeirão Preto Medical School. São Paulo University (USP)
Locations (1):
- Clinical Hospital of Ribeirao Preto, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Background] Blot SI, Depuydt P, Annemans L, Benoit D, Hoste E, De Waele JJ, Decruyenaere J, Vogelaers D, Colardyn F, Vandewoude KH. Clinical and economic outcomes in critically ill patients with nosocomial catheter-related bloodstream infections. Clin Infect Dis. 2005 Dec 1;41(11):1591-8. doi: 10.1086/497833. Epub 2005 Oct 25. PMID 16267731
- [Background] Walshe LJ, Malak SF, Eagan J, Sepkowitz KA. Complication rates among cancer patients with peripherally inserted central catheters. J Clin Oncol. 2002 Aug 1;20(15):3276-81. doi: 10.1200/JCO.2002.11.135. PMID 12149302
- [Background] Pittiruti M, Hamilton H, Biffi R, MacFie J, Pertkiewicz M; ESPEN. ESPEN Guidelines on Parenteral Nutrition: central venous catheters (access, care, diagnosis and therapy of complications). Clin Nutr. 2009 Aug;28(4):365-77. doi: 10.1016/j.clnu.2009.03.015. Epub 2009 May 21. PMID 19464090
- [Background] Maiefski M, Rupp ME, Hermsen ED. Ethanol lock technique: review of the literature. Infect Control Hosp Epidemiol. 2009 Nov;30(11):1096-108. doi: 10.1086/606162. PMID 19803767
- [Background] Safdar N, Maki DG. Inflammation at the insertion site is not predictive of catheter-related bloodstream infection with short-term, noncuffed central venous catheters. Crit Care Med. 2002 Dec;30(12):2632-5. doi: 10.1097/00003246-200212000-00003. PMID 12483050
- [Background] Raad I, Hanna H, Maki D. Intravascular catheter-related infections: advances in diagnosis, prevention, and management. Lancet Infect Dis. 2007 Oct;7(10):645-57. doi: 10.1016/S1473-3099(07)70235-9. PMID 17897607
- [Background] Cheung E, Baerlocher MO, Asch M, Myers A. Venous access: a practical review for 2009. Can Fam Physician. 2009 May;55(5):494-6. No abstract available. PMID 19439704
- [Background] Pires DPL, Afonso JC, Chaves FAB. A termometria nos séculos XIX e XX. Rev. Bras. Ensino Fís. 28(1): 101-114, 2006
- See also: Record in the Brazilian Committee of Ethics in Research — http://portal2.saude.gov.br/sisnep/pesquisador/extrato_projeto.cfm?CODIGO=377337